CLINICAL TRIAL: NCT00568711
Title: Controlled Trial: 5-day Course of Rifampin Versus Doxycycline for the Treatment of Mild to Moderate Scrub Typhus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dong-Min Kim (Other)
Responsible Party: Sponsor-Investigator, Dong-Min Kim, Chosun University Hospital, Chosun University Hospital
Organization: Chosun University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB043-31; IRB043-31
Record Dates: First submitted 2007-12-05; First posted 2007-12-06 (Estimated); Last update posted 2019-02-08 (Actual); Status verified 2019-02

CONDITIONS: Scrub Typhus
Keywords: Doxycycline,; Rifampin; Scrub typhus.
MeSH Terms: conditions — Scrub Typhus | interventions — Doxycycline; Rifampin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): a 5-day course of daily 200-mg doses of doxycycline
  Interventions: Drug: doxycycline
- 2 (Active Comparator): a 5-day course of daily 600-mg doses of rifampin
  Interventions: Drug: rifampin

INTERVENTIONS:
Drug: doxycycline — a 5-day course of 100 mg bid doses of doxycycline
  Arms: 1
Drug: rifampin — a 5-day course of daily 600-mg doses of rifampin
  Arms: 2

SUMMARY:
New antibiotics are required to have not only the antibacterial activity against doxycyline-resistant O. tsutsugamushi but also lower risk for resistance or any cross-resistance to others.

In this prospective, open-label, randomized trial, we enroll patients with mild-to-moderate scrub typhus. We compared the efficacy and safety of a 5-day rifampin therapy with those of a 5-day doxycycline therapy at Chosun University Hospital, or one of its two community-based affiliated hospitals which are all located in southwestern Korea between 2006 and 2009.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria were:

* Adults aged 18 years or older
* A fever of higher than 37.5°C
* The concurrent presence of eschar or a maculopapular skin rash; and the clear presence of more than two symptoms such as headache, malaise, myalgia, coughing, nausea and abdominal discomfort.
* Patients were hospitalized at Chosun University Hospital in Kwangju, Korea or one of its two community-based affiliated hospitals which are all located in southwestern Korea between 2006 and 2009.

Exclusion Criteria:

The exclusion criteria were:

* An inability to take oral medications
* Pregnancy
* Hypersensitivity to the trial drugs
* Previous drug therapy with potential antirickettsial activity (e.g., rifampicin, chloramphenicol, macrolides, fluoroquinolones or tetracyclines) within 48 h prior to admission
* Severe scrub typhus (shock requiring vasopressor therapy for more than one hour
* A stuporous or comatose level of consciousness
* Respiratory failure requiring mechanical ventilation or renal failure requiring immediate dialysis) (4, 10).
* For the differential diagnosis of scrub typhus from other diseases with similar symptoms (e.g., murine typhus, leptospirosis, hemorrhagic fever with renal syndrome and systemic lupus erythematosus), patients underwent diagnostic tests. We thus excluded patients with concurrent infections who had the risk of causing different outcomes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 476 (Actual)
Dates: Start 2006-09 (Actual); Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
The primary end point was the fever clearance time | 4 years

SECONDARY OUTCOMES:
The secondary end point was evaluated according to the following definitions. "Cure ", "Failure", "Relapse" | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Namsoo Cho, Study Director — Director of Chosun University Hospital
Locations (1):
- Chosun University Hospital, Gwangju, Jeollanam-do, South Korea

REFERENCES:
- [Derived] Kim YS, Kim DM, Yoon NR, Jang MS, Kim CM. Effects of Rifampin and Doxycycline Treatments in Patients With Uncomplicated Scrub Typhus: An Open-Label, Randomized, Controlled Trial. Clin Infect Dis. 2018 Aug 1;67(4):600-605. doi: 10.1093/cid/ciy130. PMID 29462266